CLINICAL TRIAL: NCT01176370
Title: A Prospective Study to Assess the Safety and Indications of Performance of the C-Pulse™ System in Relieving Heart Failure Symptoms in Patients With ACC/AHA Stage C, NYHA Class III-ambulatory Class IV Heart Failure.
Brief Title: C-Pulse Implantable Counterpulsation Pump (ICP) - A Heart Assist Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment for this study was stopped following approval of the C-Pulse System pivotal study IDE.This decision was not based on any safety concerns.
Sponsor: Nuwellis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 02977 Rev - B
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Device; Implantable; Active; Class III and Class IV; Counterpulsation
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Intervention Model Description: All enrolled/consented subjects receive study device: C-Pulse™ (Implantable Counterpulsation Therapy).
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implantable Counterpulsation Therapy (Experimental): The study is a single arm study with up to 20 patients enrolled and implanted with implantable counterpulsation. Patients that meet eligibility will be enrolled and implanted into the treatment arm of the study. There is not a control arm in this feasibility study.
  Interventions: Device: C-Pulse™ (Implantable Counterpulsation Therapy)

INTERVENTIONS:
Device: C-Pulse™ (Implantable Counterpulsation Therapy) — C-Pulse System is an implantable, non-blood contacting, non-obligatory, heart assist device.
  Other Names: C-Pulse; Implantable Counterpulsation Pump; Heart Assist System; Sunshine Heart C-Pulse ICP

SUMMARY:
The C-Pulse Study is evaluating the safety and performance of a new product for the treatment of heart failure. The product is designed to help reduce the symptoms of heart failure and help patients function better with daily activities. The study evaluates multiple measures of heart function and whether the patient's quality of life has been improved since the device implant. The patient will have several visits after the device implant to assess how well they are doing and to monitor any safety concerns.

DETAILED DESCRIPTION:
Sunshine Heart Inc. is sponsoring a prospective trial to assess the safety and provide indications for performance of the Sunshine Heart C-PulseTM System ("C-Pulse™").

The current need is for a counterpulsation device or method that is effective enough to make its application appealing as a long-term implant to a large number of patients and physicians. It must be simple and safe, with a straight-forward implant procedure, and with long-term measurable patient benefits. Further, it would be advantageous for the counterpulsation device to be smaller, easier to insert, ambulatory, disconnectable, and not in the bloodstream. Such a device may be more readily adopted by a wider group of cardiologists and surgeons, and be suitable for a wider group of people in NYHA Class III or IV heart failure. It is important to point out that a counterpulsation device is aimed to augment native heart function and is fundamentally different from total artificial hearts, left ventricular assist devices and heart transplants which are meant to be a total replacement or an alternative to the native heart. Thus, the counterpulsation device is considered non-obligatory and not life-supporting.

Sunshine Heart, Inc has proposed C-Pulse™, a novel ambulatory, non-obligatory, non-blood contacting extra-ascending aortic counterpulsation system. The C-Pulse™ System is designed to be implanted without the need for cardiopulmonary bypass or extensive dissection, to be able to be activated immediately, to augment heart function in a safe manner and to provide sustained relief from heart failure symptoms. It can be turned off safely, and similarly, in failure modes, is considered to have an associated low risk of death or disability, other than the recurrence of heart failure symptoms. C-Pulse™ is not an alternative to the heart, it is an augmentation device, and it does not preclude the use of therapies that provide full circulatory support such as heart transplantation or LVADs.

The C-Pulse™ System consists of a counterpulsation Cuff secured around the outside of the ascending aorta, the main blood vessel out of the heart. The Cuff and a heart signal sensing wire are attached to an external driver. The external Driver inflates and deflates the Cuff in sequence with the ECG signal to assist heart function and improve the pumping capacity of the heart. The Cuff deflects the aorta in a "thumb-printing" manner which has been optimized to minimize aortic wall strain and maximize blood volume displacement per beat. The C-Pulse™ System is non-blood contacting, simple to insert, and can be turned on and off as required; all natural blood pathways are maintained - there is no exposure of foreign material to the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* Patient has ACC/AHA Stage C heart failure and remains in NYHA Class III - ambulatory Class IV despite optimal medical therapy.
* ACE inhibitor or ARB (Angiotensin Receptor Blocks) at least 30 days preceding implant or nitrate/hydralazine at the investigators discretion
* Beta-blocker for at least 90 days and stable for 30 days preceding implant
* Patient has left ventricular ejection fraction (LVEF) ≤ 35%
* Patient has had Cardiac Resynchronization Therapy (CRT) for at least 90 days prior to enrollment or is not indicated for a CRT device
* Patient has had an implanted cardio-defibrillator (ICD) at least 30 days prior to enrollment or is not indicated for ICD implantation.
* Patient is at least 18 years of age and not older than 75 years
* Patient six minute hall walk assessment between 100-350 meters
* Patient understands the nature of the procedure, is willing to comply with associated follow-up evaluations, and provide written informed consent prior to the procedure

Exclusion Criteria:

* Patient has any evidence of:

  * Ascending aortic calcification on posterior-anterior or lateral chest x-ray at initial screening OR
  * Atherosclerotic ascending aortic disease, specifically intimal thickening greater than 3mm or mobile atheroma (moderate) or mural calcification (severe) as detected by CT scan or echocardiography (Echo)
* Patient has ascending aorto-coronary artery bypass grafts, history of aortic dissection, Marfans disease or other connective tissue disorder or has had an aortic root replacement
* Patient aorta not conforming to specified dimensional constraints defined by CT scan, most specifically mid ascending aortic outside diameter less than 29mm or greater than 40mm
* Patient has severe mitral valve incompetence, grade 4+
* Patient has moderate to severe aortic valve incompetence, grade 2-4+
* Patient has systolic blood pressure less than 90 or greater than 140 mmHg
* Patient has a Serum Sodium less than 130 mEq/L
* Patient has a Estimated Glomerular Filtration Rate (GFR) less than 40 ml/min/1.73m2
* Patient has any two of three of Bilirubin, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) greater than three times upper limit of normal
* Patient has a serum Albumin less than 3.0 g/dL
* Patient has Body Mass Index (BMI) less than 18 or greater than 40 kg/m2
* Patient has any active infection
* Patient has had a myocardial infarction (MI), stroke, transient ischemic attack (TIA), cardiac or other major surgery, in the 90 days prior to enrollment
* Patient has severe Chronic Obstructive Pulmonary Disease (COPD) as evidenced by Forces Expiratory Volume (FEV1) less than or equal to 0.9 L/min
* Patient requires a concomitant surgical procedure [i.e. coronary artery bypass graft (CABG), Valve repair]
* Patient is supported with a left ventricular assist device or IABP
* Severe Right Heart Dysfunction with systemic venous congestion evidenced by clinical signs/symptoms such as Central Venous Pressure (CVP) ≥ 20 mmHg, Cardiac Index (CI) < 2.0 l/min./m2, elevated liver function tests beyond three time the upper limit of normal and presence of ascites
* Patient has reversible causes of heart failure that may be remedied by conventional surgery or other intervention
* Patient is pregnant; Note: Negative pregnancy test required in all women of child bearing potential
* Patient has any other condition that, in the opinion of the investigators, would disqualify the patient for inclusion in the study, limits survival to less than one year, or not permit valid consideration
* Patient is currently enrolled or has participated in the last 30 days in another therapeutic or interventional clinical study that is likely to confound study results
* Patient has symptomatic Carotid artery disease or asymptomatic disease with a stenosis greater than 70%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-06-21 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Percent of Patients with a Device-Related Adverse Event | Through 6 months
  The primary safety endpoint is the composite device-related adverse event rate as defined by the percent of patients who experience at least one device-related adverse events out of the total number of patients.
Quality of Life (QOL) | 6 months
  improvement from baseline to 6-months post-implant. QOL as measured by the Minnesota Living with Heart Failure (MLWHF) questionnaire.
New York Heart Association (NYHA) Classification | 6 months
  improvement from baseline to 6-months post-implant. Participant NYHA Classification at 6 month follow up. The NYHA Classification involved 4 classes.
  I No limitation of physical activity II Slight limitation of physical activity III Marked limitation of physical activity IV Unable to carry on any physical activity without discomfort
Improvement in 6 Minute Walk Test (6MWT) | 6 months
  improvement from baseline to 6-months post-implant. The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.

SECONDARY OUTCOMES:
Further assess risks and benefits | 5-years
  Endpoints consistent with primary outcomes will be evaluated at additional time points and device failure rate and adverse event rates will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Renzo Cecere, MD, Principal Investigator — McGill University Health Centre, Royal Victoria Hospital
Locations (1):
- McGill University Health Centre - Royal Victoria Hospital, Montreal, Quebec, Canada